CLINICAL TRIAL: NCT03601455
Title: Phase II Study of Radiation Therapy and Anti-PD-L1 Checkpoint Inhibitor (Durvalumab) With or Without Anti-CTLA-4 Inhibition (Tremelimumab) in Patients With Unresectable, Locally Advanced, or Metastatic Urothelial Bladder Cancer That Are Ineligible or Refusing Chemotherapy
Brief Title: Radiation Therapy and Durvalumab With or Without Tremelimumab in Treating Participants With Unresectable, Locally Advanced, or Metastatic Bladder Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-001894; NCI-2018-01415 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-001894 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Bladder Urothelial Carcinoma; Stage IV Bladder Cancer AJCC v8; Stage IVA Bladder Cancer AJCC v8; Stage IVB Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab; Immunoglobulin G; Disulfides; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Regimen A (radiation therapy and durvalumab) (Experimental): Participants receive durvalumab IV over 60 minutes on day 1. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity. Participants also undergo EBRT for 5 fractions beginning on day 8 of course 1.
  Interventions: Biological: Durvalumab; Radiation: External Beam Radiation Therapy
- Regimen B (radiation therapy, durvalumab, tremelimumab) (Experimental): Participants receive tremelimumab IV over 60 minutes on day 1 for up to 2 courses and durvalumab IV over 60 minutes on day 1. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression of unacceptable toxicity. Participants also receive undergo EBRT for 5 fractions beginning on day 8 of course 1.
  Interventions: Biological: Durvalumab; Radiation: External Beam Radiation Therapy; Biological: Tremelimumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab
  Arms: Regimen B (radiation therapy, durvalumab, tremelimumab)

SUMMARY:
This phase II trial studies the side effects and how well radiation therapy and durvalumab with or without tremelimumab work in treating participants with bladder cancer that cannot be removed by surgery, has spread to nearby tissue or lymph nodes, or that has spread to other parts of the body. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Monoclonal antibodies, such as durvalumab and tremelimumab, may interfere with the ability of tumor cells to grow and spread. It is not yet known whether giving radiation therapy and durvalumab with or without tremelimumab will work better in treating participants with bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile of radiation therapy (RT) and durvalumab with or without tremelimumab. (Safety lead-in cohort) II. To determine the median progression-free survival with RT and durvalumab with or without tremelimumab. (Expansion cohort)

SECONDARY OBJECTIVES:

I. To assess the efficacy of RT and durvalumab with or without tremelimumab in terms of local control of irradiated bladder tumor.

II. To assess the efficacy of RT and durvalumab with or without tremelimumab in terms of pathologic complete response (CR) rate of irradiated bladder tumor.

III. To assess the efficacy of RT and durvalumab with or without tremelimumab in terms overall response rate.

IV. To assess the efficacy of RT and durvalumab with or without tremelimumab in terms of abscopal response rate.

V. To assess the efficacy of RT and durvalumab with or without tremelimumab in terms of duration of response.

VI. To assess the efficacy of RT and durvalumab with or without tremelimumab in terms of disease specific survival.

VII. To assess the efficacy of RT and durvalumab with or without tremelimumab in terms of overall survival.

VIII. To further determine the safety and tolerability of RT + durvalumab with or without tremelimumab (expansion cohorts).

EXPLORATORY OBJECTIVES:

I. To explore the immunologic changes associated with the combination of durvalumab and RT +/- tremelimumab.

OUTLINE: Participants are randomized to 1 of 2 regimens.

REGIMEN A: Participants receive durvalumab intravenously (IV) over 60 minutes on day 1. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity. Participants also undergo external beam radiation therapy (EBRT) for 5 fractions beginning on day 8 of course 1.

REGIMEN B:

Participants receive tremelimumab IV over 60 minutes on day 1 for up to 2 courses and durvalumab IV over 60 minutes on day 1. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression of unacceptable toxicity. Participants also receive undergo EBRT for 5 fractions beginning on day 8 of course 1.

After completion of study treatment, participants are followed up at 8 weeks and then every 12 and 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* cT2 - T4 or metastatic (N+ or M+) urothelial bladder cancer. Mixed histologies with predominant urothelial pattern are allowed. Patients with localized disease must either refuse cystectomy or be deemed not ideal cystectomy candidates.
* If metastatic disease present patients must have an intact, symptomatic bladder tumor, appropriate for palliative RT to the bladder.
* Measurable metastatic disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria. Thus, patients with metastatic disease must have at least 1 lesion, not previously irradiated, that can be accurately measured at baseline as >= 10 mm in the longest diameter (except lymph nodes which must have a short axis >= 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and that is suitable for accurate repeated measurement as per RECIST v1.1 guidelines.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1/
* Life expectancy of >= 12 weeks.
* Patients must be ineligible for or refuse cisplatin-based chemotherapy. Cisplatin ineligibility is defined as meeting 1 of the following criteria:

  * Creatinine clearance (calculated or measured) < 60 mL/min
  * Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 audiometric hearing loss
  * CTCAE grade 2 or higher peripheral neuropathy
  * New York Heart Association class III heart failure
  * Any other criteria deemed by the investigator to make the patient unsuitable for cisplatin-based chemotherapy

    * Note: The reason for cisplatin ineligibility must be documented. Patients may refuse cisplatin-based chemotherapy after an informed discussion of the risks and benefits, and the reason for refusal must be documented.
* Subjects must consent to provide an archived tumor specimen from within 12 months prior to study entry (ie, from subject signing consent to participate in the study) for immunologic characterization. If not available, subjects should have at least 1 lesion amenable to biopsy and consent to provide a pre-treatment fresh biopsy. Tumor lesions used for biopsy should not be lesions used as target lesions. Additional archival tissue from beyond 12 months prior to study entry is also requested, if available, to support exploratory analyses.
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (>= 1500 per mm^3)
* Platelet count >= 100 x 10^9/L (>= 100,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert?s syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be =< 5 x ULN
* Serum creatinine clearance (CL) > 30 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance.
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: >= 60 years old and no menses for 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visit and examinations and follow-up.

Exclusion Criteria:

* ECOG PS 2 or higher.
* Prior cystectomy or definitive RT to the bladder.
* History of autoimmune disease, including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegner?s granulomatosis, Sjogren?s syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], celiac disease, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Subjects with childhood atopy or asthma, vitiligo, alopecia, Hashimoto syndrome, Grave?s disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone are not excluded.
  * Patients with controlled type 1 diabetes mellitus on a stable dose of insulin regimen are not excluded.
  * Any chronic skin condition that does not require systemic therapy are not excluded.
  * Patients without active autoimmune disease in the last 5 years may be included after consultation with the study physician.
* Patients with human immunodeficiency virus (HIV), active hepatitis B (HBV) or active hepatitis C (HCV)

  * Patients with past HBV infection or resolved HBV infection, defined as the presence of hepatitis B core antibody (HBc Ab) and absence of hepatitis B surface antigen (HBsAg) are eligible. HBV deoxyribonucleic acid (DNA) must be obtained in these patients prior to day 1 of therapy, but detection of HBV DNA in these patients will not exclude study participation.
  * Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
* Previous investigational product (IP) assignment in the present study.
* Current enrollment/participation in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study.
* Prior radiation therapy to the abdomen or pelvis, including radiation therapy to the bladder, prostate, or rectum.
* Any concurrent systemic chemotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (i.e. hormonal replacement therapy) is acceptable. Prior systemic therapies are allowed with a washout period of >= 45 days.
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP. Note biopsy and transurethral resection of the bladder tumor (TURBT) of the primary tumor is acceptable.
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 3 years before the first dose of study drug and of low potential risk for recurrence.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ >> (Optional criteria that are dependent on the patient population under investigation.)

    * Note: Patients with incidental finding of early stage prostate cancer will not be eligible.
* QT interval corrected for heart rate using Fridericia?s formula (QTcF) >= 470 ms calculated. Any clinically significant abnormalities detected require triplicate electrocardiography (ECG) results and a mean QT interval corrected for heart rate using Fridericia?s formula (QTcF) >= 470 ms calculated from 3 ECGs).
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* History of hypersensitivity to durvalumab, tremelimumab, or any excipient.
* History of hypersensitivity to the combination therapy of durvalumab and tremelimumab.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and tuberculosis [TB] testing in line with local practice).
* History of leptomeningeal carcinomatosis.
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Brain metastases or spinal cord compression unless the patient?s condition is stable (asymptomatic, no evidence of new or emerging brain metastases) and off steroids for at least 14 days prior to the start of study treatment. Following radiotherapy and/or surgery, patients with suspected brain metastases at screening should have a magnetic resonance imaging (MRI)(preferred)/CT, preferably with IV contrast.
* Subjects with uncontrolled seizures.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 4.03 criteria (Safety lead-in cohort) | Up to 90 days after last dose of investigation product
  Observed toxicities will be tabulated using frequencies and percentages based on the CTCAE v 4.03.
Progression- free survival (PFS) assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 (Expansion cohort) | From the first day of the treatment to the first occurrence of disease progression or death, assessed up to 3 years
  PFS will be estimated in each study arm by Kaplan-Meier estimate, where PFS is a composite endpoint based on radiologic progression, clinical deterioration or death. A log rank test will be used to test if there is significant difference in PFS between two arms. PFS will be also estimated for localized patients and metastatic patients separately within each arm and stratified log rank test will be used as well.

SECONDARY OUTCOMES:
Local control at the primary irradiate site determined by RECIST v 1.1 | Up to 3 years
  The stratified Kaplan Meier method will be used to describe local control for each arm along with their median.
Pathologic complete rate (CR) of primary irradiated tumor | Up to 3 years
  The point estimate and its 95% confidence interval will be obtained for the pathologic CR rate of the primary irradiated tumor for each arm and for localized patients and metastatic patients separately within each arm. A two-sample proportion test will be used to test if there is significant difference in pathologic CR (pCR) rates between two arms and the CochranMantel-Haenszel test will be used when accounting for the stratified design.
Overall response rate (ORR) defined as the number (%) of patients with at least 1 visit response of CR or partial response (PR) determined by RECIST v 1.1 | Up to 3 years
  The point estimate and its 95% confidence interval of ORR will be obtained by arm and for localized patients and metastatic patients separately within each arm. A two-sample proportion test will be used to test if there is significant difference in ORR rates between two arms and the Cochran-Mantel-Haenszel test will be used when accounting for the stratified design.
Abscopal response (in patients with metastatic disease) determined by RECIST v 1.1 with response (PR and CR) sites away from the primary irradiated tumor | Up to 3 years
  The point estimate and its 95% confidence interval will be obtained by arm and for localized patients and metastatic patients separately within each arm. Furthermore, a two-sample proportion test will be used to test if there is significant difference between two arms and the Cochran-Mantel-Haenszel test will be used when accounting for the stratified design.
Duration of response | From date of the first documented response until the first date of documented progression or death, assessed up to 3 years
  The stratified Kaplan Meier method will be used to describe the duration of response for each arm along with their median.
Disease-specific survival | From the date of randomization to the date of death related to treatment and/or disease determined, assessed up to 3 years
  The stratified Kaplan Meier method will be used to describe disease-specific survival for each arm along with their median.
Overall survival | From the date of randomization to the date of to the date of death due to any cause, assessed up to 3 years
  The stratified Kaplan Meier method will be used to describe overall survival for each arm along with their median.
Incidence of adverse events assessed by National Cancer Institute CTCAE v4.0 | Up to 3 years
  Will be summarized according to the subjects? baseline grade and maximum grade for each cycle of therapy.

OTHER OUTCOMES:
Immune cell subsets and PD-L1 assessed by immunohistochemistry in tumor biopsies | Up to 3 years
  Will be summarized by descriptive statistics. Frequency distribution and percentage will be used to summarize PD-L1 expression at baseline and at time of progression.
Gene signature biomarker | Baseline
  Two-sample Wilcoxon tests to compare patients who achieve uncoupling and those who do not for each arm. Adjusted P values controlling for false discovery rate (Benjamini and Hochberg method) will be derived. For genes or signatures that emerge as significantly associated with response, logistic regression models will be used to assess their independent association with response. Association of gene expression levels at baseline and PFS will be explored using the Cox proportional hazards regression model. Hierarchical clustering superimposed with response status, relevant baseline or prognostic characteristics or experimental factors will be performed using Spearman correlation and complete linkage to visualize the discriminating power of the immune gene expression and the correlative structure among the genes and the samples.
Circulating immune cell subsets assessed via flow cytometry in peripheral blood mononuclear cell | Up to 3 years
  Established flow cytometry panels will examine B cell and T cell populations. Immune cell quantification will be summarized by changes from baseline, on-, to post-treatment using descriptive statistics. Furthermore, paired Wilcoxon signed-rank test will be applied to test the pre-on, and on-post treatment changes. When available, immune cells digested from resected tumor tissues will also be assessed by flow cytometry.
Change in circulating and tumor-infiltrating T-cell receptor (TCR) repertoire | Baseline up to 3 years
  Will be assessed by calculating the number of unique clonotypes, read depth and Shannon diversity index. Repertoire overlap and change between sequencing experiments will be measured using Baroni-Urbani and Buser overlap index and Morisita?s distance, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Chang, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States